CLINICAL TRIAL: NCT06970366
Title: Cryotherapy and Muscle Function: Assessing Injury Risk in Immediate Return-to-Play Scenarios
Brief Title: Cryotherapy on Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Berna Cagla Balkisli, Assist. Prof., Okan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OkanUNI
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cold; Cryotherapy; Cryotherapy Effect; Muscle Activity; EMG
Keywords: cryotherapy; muscle activity
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold pack group (Experimental): Participants in this group will receive a standard cold pack application to the target muscle area while in a relaxed position. The cold pack, maintained at a temperature between 0-5°C, will be applied directly over the skin with a thin cloth barrier to prevent frostbite. The application will last for 10 minutes.
  Interventions: Other: Cold pack application
- Cold spray group (Active Comparator): Participants in this group will receive a cold spray application to the target muscle area while in a relaxed position. A commercially available vapocoolant spray (e.g., ethyl chloride or similar) will be applied from a distance of approximately 20 cm in a sweeping motion for 5-10 seconds until the skin reaches a visible cooling effect without causing frostbite or discomfort.
  Interventions: Other: Cold spray application

INTERVENTIONS:
Other: Cold pack application — Cold pack application
  Arms: Cold pack group
Other: Cold spray application — Cold spray application
  Arms: Cold spray group

SUMMARY:
On-field sports injuries are a common issue that significantly impacts athletes' performance and overall health. In team sports such as football, basketball, and volleyball, muscle and joint injuries are particularly frequent. Cryotherapy, including cold pack and cold spray applications, is widely used in the acute management of such injuries due to its practicality and rapid application. It is effective in reducing pain and edema by constricting blood vessels and slowing neural activity. While its analgesic effects are well-known, some studies suggest cryotherapy may also influence balance and proprioception. This study aims to investigate the acute effects of cryotherapy (cold pack and spray) on muscle mechanical properties, muscle strength, pain and EMG activity in healthy individuals.

A randomized, controlled experimental study will be conducted on healthy participants. Subjects will be divided into two groups: cold pack application and cold spray application. Quadriceps muscle mechanical properties will be assessed using a Myoton device; muscle strength will be evaluated via dynamometry, and muscle activity will be evaluated via electromyographic (EMG) device- NeuroTrac® MyoPlus 2. Each participant will be evaluated at four time points: baseline (pre-intervention), immediately after the intervention, 3 minutes post-intervention, and 5 minutes post-intervention. The effects of each modality will be compared both within and between groups to assess the short-term physiological changes induced by cryotherapy.

ELIGIBILITY:
Inclusion Criteria:

* being male
* aging 18-25
* having no history of cardiovascular or peripheral vascular disease, diabetes mellitus, neuromuscular pathology, peripheral neuropathy, lower extremity pain, or previous lower extremity surgery
* being volunteer

Exclusion Criteria:

* having a history of insensitivity to local heat or cold

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Muscle Properties | from the application (baseline), immediately after the application, 3 minutes post-application, and to 5 minutes post-application.
  The assessment of muscle mechanical properties will be performed using the MyotonPRO device. Measurements will be taken bilaterally from the quadriceps muscle, specifically targeting the knee extensors.
Muscle strength | from the application (baseline), immediately after the application, 3 minutes post-application, and to 5 minutes post-application.
  The isometric muscle strength of the participants' dominant quadriceps muscle will be measured using a dynamometer. Muscle strength assessments will be performed with a calibrated Lafayette dynamometer (model 01163; Lafayette Instrument Company, Lafayette, IN, USA). Participants will receive verbal instructions about the procedure prior to testing. During the assessment, care will be taken to ensure that the device does not slip, that appropriate force is applied, that no compensatory movements occur in the tested extremity or other body parts, and that weakness is not masked by body positioning. For knee extensor evaluation, participants will be seated with their hands crossed over their shoulders, hips flexed at 90°, and knees locked at 60° of extension.
Muscle activity | from the application (baseline), immediately after the application, 3 minutes post-application, and to 5 minutes post-application.
  The EMG activity of the participants' dominant quadriceps muscle will be measured using a surface electromyography (EMG) device. For this assessment, the NeuroTrac® MyoPlus 2 dual-channel EMG ETS device (Verity Medical Ltd., UK) will be used. The device will be connected to a computer via dedicated software. To measure muscle activity, 32 mm diameter, circular, adhesive silver-silver chloride (Ag-AgCl) electrodes will be used. Three electrodes will be prepared individually for each participant. Prior to placement, the skin area where the surface electrodes will be attached will be cleaned with an alcohol wipe to reduce skin impedance. A reference electrode will be placed on the leg to eliminate external interference, while the active electrodes will be positioned directly over the target muscle.

SECONDARY OUTCOMES:
Pressure pain threshold | from the application (baseline), immediately after the application, 3 minutes post-application, and to 5 minutes post-application.
  The pressure pain threshold (PPT) of the dominant quadriceps muscle will be assessed using a digital pressure algometer. The algometer is equipped with a flat circular rubber-tipped probe (1 cm²) and will be applied perpendicularly to the skin over the quadriceps muscle belly. The probe will be pressed gradually at a constant rate (approximately 1 kg/cm² per second) until the participant reports the sensation of pressure turning into pain. The corresponding force value will be recorded as the PPT. Each participant will receive verbal instructions prior to the test, and the measurement site will be marked to ensure consistency across repeated measures. The assessment will be performed in a seated and relaxed position, with care taken to avoid muscle contraction or movement during the measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cryotherapy for acute musculoskeletal injuries: a systematic review and meta-analysis.